CLINICAL TRIAL: NCT00525330
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of KRP-104 in Patients With Type 2 Diabetes Inadequately Controlled on Metformin Alone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ActivX Biosciences, Inc. (Industry)
Collaborators: Kyorin Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0104-003
Record Dates: First submitted 2007-09-03; First posted 2007-09-05 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- KRP-104 120 mg QD (Experimental)
  Interventions: Drug: KRP-104 QD Drug: Placebo Drug: Metformin
- KRP-104 60 mg BID (Experimental)
  Interventions: Drug: KRP-104 BID Drug: Placebo Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Drug: Metformin

INTERVENTIONS:
Drug: KRP-104 QD Drug: Placebo Drug: Metformin — KRP-104 120 mg: KRP-104 two 50 mg tablets and two 10 mg tablets 15 to 30 minutes before morning meal and 2 placebo tablets 15 to 30 minutes before evening meal
  Arms: KRP-104 120 mg QD
Drug: Placebo Drug: Metformin — Two tablets 15 to 30 minutes before each meal, morning and evening.
  Arms: Placebo
Drug: KRP-104 BID Drug: Placebo Drug: Metformin — KRP-104 60 mg: KRP-104 one 50 mg tablet plus one 10 mg tablet 15 to 30 minutes before each meal, morning and evening.
  Arms: KRP-104 60 mg BID

SUMMARY:
To assess the safety and efficacy of chronic therapy with KRP-104, a novel DPP-IV inhibitor, in patients with Type 2 Diabetes on stable metformin therapy. In addition, an estimate of how much of the HbA1c response is attributable to nocturnal coverage will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years, inclusive;
2. Males and females of non-childbearing potential;
3. Diagnosis of type 2 diabetes mellitus according; and
4. On a stable dose of metformin monotherapy at randomization (can be on other oral therapies or naive at study entry

Exclusion Criteria:

1. History of type 1 diabetes mellitus or history of diabetic ketoacidosis or persistent hypoglycemia;
2. History or presence of alcoholism or drug abuse
3. Typical consumption of ≥10 drinks of alcohol weekly;
4. Presence of any of the following conditions:

   * Significant renal impairment (glomerular filtration rate <60 mL/min [to be calculated by the central laboratory]);
   * Diabetic retinopathy;
   * Diabetic gastroparesis;
   * Active liver disease (other than asymptomatic nonalcoholic fatty liver disease), cirrhosis, or symptomatic gallbladder disease;
5. Uncontrolled high blood pressure;
6. History or evidence of cardiovascular or pulmonary disease
7. Must meet other laboratory and Medical History clinical criteria. Please contact recruitment center for referrals

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial is to demonstrate the hemoglobin A1c (HbA1c)-lowering effects of KRP-104 in patients with type 2 diabetes inadequately controlled on metformin alone. | 12-weeks

SECONDARY OUTCOMES:
To assess the fasting plasma glucose (FPG)-lowering effect of KRP-104 in patients with type 2 diabetes inadequately controlled on metformin alone; | 12-weeks
To compare effects of once daily (QD) dosing versus twice daily (BID) dosing of KRP-104 on HbA1c and FPG | 12 weeks
To assess the effects of KRP-104 on post-prandial glucose dynamics and insulin sensitivity (homeostasis model index [HOMA-β]) in the setting of a Meal Tolerance Test(MTT) | 12 weeks
  Changes from pre-prandial to 2-hour post-prandial glucose, active GLP-1, insulin summarized by treatment group from Week 0 to Week 5 and Week 12. Percent change in 2-hour post-prandial glucose summarized by treatment group from Week 0 to Week 5 and Week 12.
To assess the safety and tolerability of KRP-104; | Daily for 12 weeks to 2 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Orloff, Study Chair — Medpace, Inc.; Tufail Syed, Study Chair — Medpace India
Locations (1):
- San Diego, California, United States